CLINICAL TRIAL: NCT02298985
Title: Curcumin as add-on to Antipsychotic Treatment in Chronic Schizophrenia Patients: A Randomized, Double-Blind, Placebo-controlled Study
Brief Title: Curcumin Addition to Antipsychotic Treatment in Chronic Schizophrenia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Tirat Carmel Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Vladimir Lerner, Associate Professor, Beersheva Mental Health Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: VLJB-14
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Chronic Schizophrenia
Keywords: curcumin; schizophrenia; neuroprotection
MeSH Terms: conditions — Schizophrenia | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- curcumin (Active Comparator): curcumin 3 g/day for 6 months
  Interventions: Drug: Curcumin; Drug: placebo
- placebo (Placebo Comparator): curcumin 3 g/day for 6 months
  Interventions: Drug: Curcumin; Drug: placebo

INTERVENTIONS:
Drug: Curcumin — 3 g/day (3 capsules/day) for 6 months
  Other Names: placebo; regular antipsychotic medication
Drug: placebo — 3 g/day (3 capsules/day) for 6 months
  Other Names: curcumin; regular antipsychotic medication

SUMMARY:
Schizophrenia is still remained one of the disabling disorders despite progress in treatment of mental disturbances. Ten to thirty percents of patients have a little or no benefit from treatment with all kinds of antipsychotics using adequate dosages and duration. Treatment of these patients has remained a persistent public health problem since medication-resistant patients are often highly symptomatic. Curcumin is one of the main curcuminoids isolated from this perennial herb. It possesses a variety of pharmacological activities, including anti-inflammatory, antiproliferative, antioxidant, and neuroprotective effects and crosses the blood-brain barrier. The purpose of our suggested study is to examine the efficacy of curcumin as add-on the conventional antipsychotic psychopharmacotherapy in chronic schizophrenia patients.

DETAILED DESCRIPTION:
Study Design This is a 24-week, randomized, double-blind, placebo-controlled investigation of 40 chronic schizophrenia patients.

Participants Forty patients will be drawn from the patient population of Be'er Sheva Mental Health Center. Recruitment period will last over 2 years.

Patients will be required to have a primary diagnosis of chronic schizophrenia as defined in DSM-IV with predominantly persistent negative signs.

The study will commence only after approval by the local Institutional Ethics Review Board ("Helsinki Committee"). Only willing subjects and able to provide written informed consent, after receiving a comprehensive explanation of the study procedures, will be included in the study. Confidentially will be ensured by means of a number coding system, and all completed research forms will be stored in secure areas.

Procedure Patients will continue receiving their regular antipsychotic medication. The dose will be kept constant for at least 3 months prior to entry and throughout the study period. Curcumin is provided as Curcumin Forte ® (Solgar Israel SupHerb). Circumin capsules are supplied as an 1000 mg soft gelatin capsule for three daily oral administration with meals. At entry patients will receive curcuma capsules (3000 mg/day, three capsules) or placebo in identical capsules in a randomized, double blind mode for 24 weeks: 20 patients will receive curcumin, and 20 patients - placebo.

Participants will be assessed at baseline and after 4, 8, 12, 16 and 24 weeks of treatment. In a case of treatment discontinuation for 24-week of the trial, patients will be followed until end of study period.

Outcome variables will be evaluated by scoring the severity of symptoms (positive, negative, and etc.), and side effects. In addition, liver function tests and a blood cell count will be monitored at baseline and during the study.

For analyzing the results, within-subject pre- and post-treatment responses would be subject to statistical procedures to evaluate whether curcumin can ameliorate the persistent negative symptoms in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years, male or female
* DSM-IV criteria for schizophrenia.
* Ability and willingness to sign informed consent for participation in the study
* SANS (Scale of Negative Symptoms of Schizophrenia ) > 30 points
* Fixed antipsychotic dosages at least 3 months
* Steady mental state of patients at least 3 months

Exclusion Criteria:

* Current substance use disorder except nicotine dependence
* Regular use of NSAID (non-steroidal anti-inflammatory drugs)
* Cancer history
* Untreated or severe hypertension
* Poorly controlled diabetes mellitus Type I or Type II
* Chronic liver & gallbladder diseases
* Recent GERD (Gastroesophageal Reflux Disorder)
* Neurological disorders: epilepsy, stroke
* Hamilton Depression Scale Hamilton Depression Rating Scale (HAM-D-17 item) > 24 points
* Patients with a known hypersensitivity to curcumin
* Pregnant women or a woman who intends to become pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptoms Scale (PANSS) | up to 24 weeks
  baseline and every week 4 up to 24 weeks

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement (CGI-I) | up to 24 weeks
  baseline and every week 4 up to 24 weeks
Clinical Global Impression - Severity of Adverse Events (CGI-SAE) | up to 24 weeks
  baseline and every week 4 up to 24 weeks
Calgary Depression Scale for Schizophrenia (CDSS) | up to 24 weeks
  baseline and every week 4 up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lerner, MD, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (2):
- Israel (2):
  - Beersheva Mental Health Center, Beersheva
  - Tirat Carmel Mental Health Center, Tirat Carmel

REFERENCES:
- [Derived] Miodownik C, Lerner V, Kudkaeva N, Lerner PP, Pashinian A, Bersudsky Y, Eliyahu R, Kreinin A, Bergman J. Curcumin as Add-On to Antipsychotic Treatment in Patients With Chronic Schizophrenia: A Randomized, Double-Blind, Placebo-Controlled Study. Clin Neuropharmacol. 2019 Jul/Aug;42(4):117-122. doi: 10.1097/WNF.0000000000000344. PMID 31045590